CLINICAL TRIAL: NCT03587805
Title: An Open-label, Single-arm, Multi-centre, Long-term Extension Trial to Evaluate the Safety and Efficacy of Tralokinumab in Subjects With Atopic Dermatitis Who Participated in Previous Tralokinumab Clinical Trials
Brief Title: Long-term Extension Trial in Subjects With Atopic Dermatitis Who Participated in Previous Tralokinumab Trials - ECZTEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0162-1337; 2018-000746-19 (EudraCT Number); U1111-1282-4519 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tralokinumab, all subjects (Experimental): Week 0: subcutaneous (SC) injection of tralokinumab loading dose. From Week 2 up to Week 266: SC injection of tralokinumab maintenance dose. The length of treatment for each subject will depend on when they enter the trial, and on which parent trial and country they come from.
  Interventions: Drug: Tralokinumab

INTERVENTIONS:
Drug: Tralokinumab — Human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. Presented as a liquid formulation for subcutaneous injection.

SUMMARY:
The purpose of this extension trial is to evaluate the long-term safety of tralokinumab.

ELIGIBILITY:
Inclusion Criteria:

* Completed the treatment period(s) of one of the parent trials: LP0162-1325, -1326, -1334, -1339, -1341, -1342, -1343, -1346, or TRA-WEI-0015-I.
* Complied with the clinical trial protocol in the parent trial to the satisfaction of the investigator.
* Able and willing to self-administer tralokinumab treatment (or have it administered by a caregiver) at home after the initial 3 injection visits at the trial site (in this trial).
* Stable dose of emollient twice daily (or more, as needed) for at least 14 days before baseline.

Exclusion Criteria:

* Any condition that required permanent discontinuation of trial treatment in the parent trial.
* More than 26 weeks have elapsed since the subject received the last injection of investigational medicinal product (IMP) in the parent trial (to be assessed at baseline).
* Subjects who, during their participation in the parent trial, developed a serious adverse event (SAE) deemed related to tralokinumab by the investigator, which in the opinion of the investigator could indicate that continued treatment with tralokinumab may present an unreasonable safety risk for the subject.
* Subjects who, during their participation in the parent trial, developed an AE that was deemed related to tralokinumab by the investigator and led to temporary discontinuation of trial treatment, which in the opinion of the investigator could indicate that continued treatment with tralokinumab may present an unreasonable safety risk for the subject.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroid within 4 weeks prior to baseline.
* Treatment with topical phosphodiesterase 4 inhibitors or topical JAK inhibitors within 2 weeks prior to baseline.
* Clinically significant infection within 4 weeks prior to baseline.
* A helminth parasitic infection within 6 months prior to the date when informed consent is obtained.
* Tuberculosis requiring treatment within 12 months prior to screening.
* Known primary immunodeficiency disorder.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1672 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical expert, Study Director — LEO Pharma
Locations (243):
- United States (83):
  - LEO Pharma Investigational Site, Birmingham, Alabama
  - LEO Pharma Investigational Site, Mobile, Alabama
  - LEO Pharma Investigational Site, Fort Smith, Arkansas
  - LEO Pharma Investigational Site, Bakersfield, California
  - LEO Pharma Investigational Site, Beverly Hills, California
  - LEO Pharma Investigational Site, Encinitas, California
  - LEO Pharma Investigational Site, Fountain Valley, California
  - LEO Pharma Investigational Site, Fremont, California
  - LEO Pharma Investigational Site, Fullerton, California
  - LEO Pharma Investigational Site, Los Angeles, California
  - LEO Pharma Investigational Site, Newport Beach, California
  - LEO Pharma Investigational Site, Northridge, California
  - LEO Pharma Investigational Site, Palo Alto, California
  - LEO Pharma Investigational Site, San Diego, California
  - LEO Pharma Investigational Site, San Francisco, California
  - LEO Pharma Investigational Site, San Luis Obispo, California
  - LEO Pharma Investigational Site, Santa Ana, California
  - LEO Pharma Investigational Site, Santa Monica, California
  - LEO Pharma Investigational Site, New Haven, Connecticut
  - LEO Pharma Investigational Site, Clearwater, Florida
  - LEO Pharma Investigational Site, Doral, Florida
  - LEO Pharma Investigational Site, Hialeah, Florida
  - LEO Pharma Investigational Site, Miami, Florida
  - LEO Pharma Investigational Site 1, Miami, Florida
  - LEO Pharma Investigational Site 2, Miami, Florida
  - LEO Pharma Investigational Site, North Miami Beach, Florida
  - LEO Pharma Investigational Site, Orange Park, Florida
  - LEO Pharma Investigational Site, Sweetwater, Florida
  - LEO Pharma Investigational Site, Tampa, Florida
  - LEO Pharma Investigational Site, West Palm Beach, Florida
  - LEO Pharma Investigational Site, Albany, Georgia
  - LEO Pharma Investigational Site, Columbus, Georgia
  - LEO Pharma Investigational Site, Macon, Georgia
  - LEO Pharma Investigational Site, Newnan, Georgia
  - LEO Pharma Investigational Site, Savannah, Georgia
  - LEO Pharma Investigational Site, Chicago, Illinois
  - LEO Pharma Investigational Site, Clarksville, Indiana
  - LEO Pharma Investigational Site, Indianapolis, Indiana
  - LEO Pharma Investigational Site, Plainfield, Indiana
  - LEO Pharma Investigational Site, Overland Park, Kansas
  - LEO Pharma Investigational Site, Louisville, Kentucky
  - LEO Pharma Investigational Site, Baton Rouge, Louisiana
  - LEO Pharma Investigational Site, Lake Charles, Louisiana
  - LEO Pharma Investigational Site, Bangor, Maine
  - LEO Pharma Investigational Site, Boston, Massachusetts
  - LEO Pharma Investigational Site, Brighton, Massachusetts
  - LEO Pharma Investigational Site, Quincy, Massachusetts
  - LEO Pharma Investigational Site, Ann Arbor, Michigan
  - LEO Pharma Investigational Site, Detroit, Michigan
  - LEO Pharma Investigational Site, Troy, Michigan
  - LEO Pharma Investigational Site, West Bloomfield, Michigan
  - LEO Pharma Investigational Site, Ypsilanti, Michigan
  - LEO Pharma Investigational Site, Saint Joseph, Missouri
  - LEO Pharma Investigational Site, Missoula, Montana
  - LEO Pharma Investigational Site, Henderson, Nevada
  - LEO Pharma Investigational Site, East Windsor, New Jersey
  - LEO Pharma Investigational Site, Buffalo, New York
  - LEO Pharma Investigational Site, Cortland, New York
  - LEO Pharma Investigational Site, Horseheads, New York
  - LEO Pharma Investigational Site, Kew Gardens, New York
  - LEO Pharma Investigational Site, New York, New York
  - LEO Pharma Investigational Site, Raleigh, North Carolina
  - LEO Pharma Investigational Site, Bexley, Ohio
  - LEO Pharma Investigational Site, Cincinnati, Ohio
  - LEO Pharma Investigational Site, Dublin, Ohio
  - LEO Pharma Investigational Site, Fairborn, Ohio
  - LEO Pharma Investigational Site, Toledo, Ohio
  - LEO Pharma Investigational Site, Tulsa, Oklahoma
  - LEO Pharma Investigational Site, Portland, Oregon
  - LEO Pharma Investigational Site, Pittsburgh, Pennsylvania
  - LEO Pharma Investigational Site, North Charleston, South Carolina
  - LEO Pharma Investigational Site, Goodlettsville, Tennessee
  - LEO Pharma Investigational Site, Austin, Texas
  - LEO Pharma Investigational Site, Bellaire, Texas
  - LEO Pharma Investigational Site, Dallas, Texas
  - LEO Pharma Investigational Site, Frisco, Texas
  - LEO Pharma Investigational Site, Houston, Texas
  - LEO Pharma Investigational Site, Pflugerville, Texas
  - LEO Pharma Investigational Site, San Antonio, Texas
  - LEO Pharma Investigational Site, Webster, Texas
  - LEO Pharma Investigational Site, South Burlington, Vermont
  - LEO Pharma Investigational Site, Norfolk, Virginia
  - LEO Pharma Investigational Site, Morgantown, West Virginia
- Belgium (9):
  - LEO Pharma Investigational Site, Brussels
  - LEO Pharma Investigational Site, Edegem
  - LEO Pharma Investigational Site, Ghent
  - LEO Pharma Investigational Site, Herstal
  - LEO Pharma Investigational Site, Kortrijk
  - LEO Pharma Investigational Site, Leuven
  - LEO Pharma Investigational Site, Liège
  - LEO Pharma Investigational Site, Loverval
  - LEO Pharma Investigational Site, Maldegem
- Canada (27):
  - LEO Pharma Investigational Site, Calgary, Alberta
  - LEO Pharma Investigational Site, Edmonton, Alberta
  - LEO Pharma Investigational Site, Surrey, British Columbia
  - LEO Pharma Investigational Site, Vancouver, British Columbia
  - LEO Pharma Investigational Site, Winnipeg, Manitoba
  - LEO Pharma Investigational Site, Bathurst, New Brunswick
  - LEO Pharma Investigational Site, Fredericton, New Brunswick
  - LEO Pharma Investigational Site, St. John's, Newfoundland and Labrador
  - LEO Pharma Investigational Site, Halifax, Nova Scotia
  - LEO Pharma Investigational Site, Ajax, Ontario
  - LEO Pharma Investigational Site, Etobicoke, Ontario
  - LEO Pharma Investigational Site, Hamilton, Ontario
  - LEO Pharma Investigational Site, London, Ontario
  - LEO Pharma Investigational Site, Markham, Ontario
  - LEO Pharma Investigational Site, Mississauga, Ontario
  - LEO Pharma Investigational Site, North Bay, Ontario
  - LEO Pharma Investigational Site, Oakville, Ontario
  - LEO Pharma Investigational Site, Ottawa, Ontario
  - LEO Pharma Investigational Site, Peterborough, Ontario
  - LEO Pharma Investigational Site, Richmond Hill, Ontario
  - LEO Pharma Investigational Site, Toronto, Ontario
  - LEO Pharma Investigational Site, Waterloo, Ontario
  - LEO Pharma Investigational Site, Windsor, Ontario
  - LEO Pharma Investigational Site, Montreal, Quebec
  - LEO Pharma Investigational Site, Québec, Quebec
  - LEO Pharma Investigational Site, Verdun, Quebec
  - LEO Pharma Investigational Site, Saskatoon, Saskatchewan
- Czechia (5):
  - LEO Pharma Investigational Site, Karlovy Vary
  - LEO Pharma Investigational Site, Kutná Hora
  - LEO Pharma Investigational Site, Ostrava-Poruba
  - LEO Pharma Investigational Site, Pardubice
  - LEO Pharma Investigational Site, Prague
- France (14):
  - LEO Pharma Investigational Site, Marseille, Bouches-du-Rhône
  - LEO Pharma Investigational Site, Bordeaux
  - LEO Pharma Investigational Site, Dijon
  - LEO Pharma Investigational Site, Grenoble
  - LEO Pharma Investigational Site, Lille
  - LEO Pharma Investigational Site, Martigues
  - LEO Pharma Investigational Site, Mulhouse
  - LEO Pharma Investigational Site, Nice
  - LEO Pharma Investigational Site, Paris
  - LEO Pharma Investigational Site, Pierre-Bénite
  - LEO Pharma Investigational Site, Rouen
  - LEO Pharma Investigational Site, Saint-Etienne
  - LEO Pharma Investigational Site, Toulouse
  - LEO Pharma Investigational Site, Valence
- Germany (26):
  - LEO Pharma Investigational Site, Aachen
  - LEO Pharma Investigational Site, Augsburg
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Berlin
  - LEO Pharma Investigational Site, Bielefeld
  - LEO Pharma Investigational Site, Bochum
  - LEO Pharma Investigational Site, Bonn
  - LEO Pharma Investigational Site, Darmstadt
  - LEO Pharma Investigational Site, Dresden
  - LEO Pharma Investigational Site, Dülmen
  - LEO Pharma Investigational Site, Erlangen
  - LEO Pharma Investigational Site, Frankfurt am Main
  - LEO Pharma Investigational Site, Friedrichshafen
  - LEO Pharma Investigational Site, Gera
  - LEO Pharma Investigational Site, Halle
  - LEO Pharma Investigational Site, Hamburg
  - LEO Pharma Investigational Site, Hanover
  - LEO Pharma Investigational Site, Jena
  - LEO Pharma Investigational Site, Kiel
  - LEO Pharma Investigational Site, Leipzig
  - LEO Pharma Investigational Site, Mainz
  - LEO Pharma Investigational Site, München
  - LEO Pharma Investigational Site, Münster
  - LEO Pharma Investigational Site, Osnabrück
  - LEO Pharma Investigational Site, Selters
  - LEO Pharma Investigational Site, Tübingen
- Italy (5):
  - LEO Pharma Investigational Site, Brescia
  - LEO Pharma Investigational Site, Catania
  - LEO Pharma Investigational Site, L’Aquila
  - LEO Pharma Investigational Site, Roma
  - LEO Pharma Investigational Site, Rozzano
- Japan (32):
  - LEO Pharma Investigational Site, Ichikawa-shi, Chiba
  - LEO Pharma Investigational Site, Chikushino-shi, Fukuoka
  - LEO Pharma Investigational Site, Fukuoka, Fukuoka
  - LEO Pharma Investigational Site, Asahikawa, Hokkaido
  - LEO Pharma Investigational Site, Sapporo, Hokkaido
  - LEO Pharma Investigational Site, Nonoichi-shi, Ishikawa-ken
  - LEO Pharma Investigational Site, Kagoshima, Kagoshima-ken
  - LEO Pharma Investigational Site, Kawasaki-shi, Kanagawa
  - LEO Pharma Investigational Site, Yokohama, Kanagawa
  - LEO Pharma Investigational Site, Toyonaka-shi, Osaka
  - LEO Pharma Investigational Site, Koto-Ku, Tokyo
  - LEO Pharma Investigational Site, Minato-Ku, Tokyo
  - LEO Pharma Investigational Site, Setagaya-ku, Tokyo
  - LEO Pharma Investigational Site, Shinjuku-Ku, Tokyo
  - LEO Pharma Investigational Site, Chūōku
  - LEO Pharma Investigational Site, Fukuoka
  - LEO Pharma Investigational Site, Fukushima
  - LEO Pharma Investigational Site, Gifu
  - LEO Pharma Investigational Site, Hamamatsu
  - LEO Pharma Investigational Site, Hyōgo
  - LEO Pharma Investigational Site, Ichinomiya
  - LEO Pharma Investigational Site, Kagoshima
  - LEO Pharma Investigational Site, Kyoto
  - LEO Pharma Investigational Site, Morioka
  - LEO Pharma Investigational Site, Nagoya
  - LEO Pharma Investigational Site, Obihiro
  - LEO Pharma Investigational Site 2, Osaka
  - LEO Pharma Investigational Site 1, Osaka
  - LEO Pharma Investigational Site, Osaka
  - LEO Pharma Investigational Site, Shimotsuke-shi
  - LEO Pharma Investigational Site, Tokyo
  - LEO Pharma Investigational Site, Toyama
- Poland (13):
  - LEO Pharma Investigational Site, Bialystok
  - LEO Pharma Investigational Site, Bochnia
  - LEO Pharma Investigational Site, Bydgoszcz
  - LEO Pharma Investigational Site, Gdansk
  - LEO Pharma Investigational Site, Gdynia
  - LEO Pharma Investigational Site, Katowice
  - LEO Pharma Investigational Site, Krakow
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Lublin
  - LEO Pharma Investigational Site, Poznan
  - LEO Pharma Investigational Site, Rzeszów
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw
- Spain (14):
  - LEO Pharma Investigational Site, Alicante
  - LEO Pharma Investigational Site, Badalona
  - LEO Pharma Investigational Site, Barakaldo
  - LEO Pharma Investigational Site, Barcelona
  - LEO Pharma Investigational Site, Bilbao
  - LEO Pharma Investigational Site, Córdoba
  - LEO Pharma Investigational Site, Fuenlabrada
  - LEO Pharma Investigational Site, Granada
  - LEO Pharma Investigational Site, L'Hospitalet de Llobregat
  - LEO Pharma Investigational Site, Madrid
  - LEO Pharma Investigational Site, Pamplona
  - LEO Pharma Investigational Site, Pontevedra
  - LEO Pharma Investigational Site, Seville
  - LEO Pharma Investigational Site, Valencia
- United Kingdom (15):
  - LEO Pharma Investigational Site, Birmingham
  - LEO Pharma Investigational Site, Cambridge
  - LEO Pharma Investigational Site, Cottingham
  - LEO Pharma Investigational Site, Dudley
  - LEO Pharma Investigational Site, Dundee
  - LEO Pharma Investigational Site, Harlow
  - LEO Pharma Investigational Site, Harrogate
  - LEO Pharma Investigational Site, Leytonstone
  - LEO Pharma Investigational Site, London
  - LEO Pharma Investigational Site, Redhill
  - LEO Pharma Investigational Site, Salford
  - LEO Pharma Investigational Site, Sheffield
  - LEO Pharma Investigational Site, Southampton
  - LEO Pharma Investigational Site, Wakefield
  - LEO Pharma Investigational Site, Walsall

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blauvelt A, Langley RG, Lacour JP, Toth D, Laquer V, Beissert S, Wollenberg A, Herranz P, Pink AE, Peris K, Fangel S, Gjerum L, Corriveau J, Saeki H, Warren RB, Simpson E, Reich K. Long-term 2-year safety and efficacy of tralokinumab in adults with moderate-to-severe atopic dermatitis: Interim analysis of the ECZTEND open-label extension trial. J Am Acad Dermatol. 2022 Oct;87(4):815-824. doi: 10.1016/j.jaad.2022.07.019. Epub 2022 Jul 19. PMID 35863467
- [Background] Guttman-Yassky E, Kabashima K, Staumont-Salle D, Nahm WK, Pauser S, Da Rosa JC, Martel BC, Madsen DE, Ropke M, Arlert P, Steffensen L, Blauvelt A, Reich K. Targeting IL-13 with tralokinumab normalizes type 2 inflammation in atopic dermatitis both early and at 2 years. Allergy. 2024 Jun;79(6):1560-1572. doi: 10.1111/all.16108. Epub 2024 Apr 2. PMID 38563683
- [Background] Blauvelt A, Pink A, Worm M, Langley RGB, Elewski BE, Gjerum L, Guttman-Yassky E. Outcomes of COVID-19 and Vaccination in Patients With Moderate to Severe Atopic Dermatitis Treated With Tralokinumab. JAMA Dermatol. 2022 Nov 1;158(11):1327-1330. doi: 10.1001/jamadermatol.2022.3488. PMID 36223087
- [Derived] Blauvelt A, Hong HC, Katoh N, Langley RG, Laquer V, Lesiak A, Peris K, Seneschal J, Silvestre JF, Warren RB, Wollenberg A, Zirwas M, Bennike NH, Safavimanesh F, Tindberg AM, Reich K. Long-Term Safety and Efficacy of Tralokinumab in Patients with Moderate-to-Severe Atopic Dermatitis Treated for up to 6 Years: Final Results from the Open-Label Extension Trial ECZTEND. Dermatol Ther (Heidelb). 2026 Feb 5. doi: 10.1007/s13555-026-01656-7. Online ahead of print. PMID 41642555
- [Derived] Mayo T, Silverberg JI, Armstrong A, Guttman-Yassky E, Blauvelt A, Esdaile B, Kabashima K, Gooderham M, Kircik L, Schneider S, Bennike N, von Eyben R, Martel BC, Ropke MA, Katoh N, Alexis AF. Efficacy and Safety of Tralokinumab Across Racial Subgroups in Adults with Moderate-to-Severe Atopic Dermatitis: Post Hoc Analysis of Phase III Trials. Am J Clin Dermatol. 2025 Oct 21. doi: 10.1007/s40257-025-00985-1. Online ahead of print. PMID 41118053
- [Derived] Reich K, Langley RG, Salvador JFS, Staumont-Salle D, Costanzo A, Pink AE, Paller AS, Katoh N, Wollenberg A, Warren RB, Blauvelt A, Oland CB, Tindberg AM, Gjerum L, Simpson EL. Safety of tralokinumab in patients with moderate-to-severe atopic dermatitis followed for up to 4.5 years: an integrated analysis of 8 clinical trials. Br J Dermatol. 2025 Aug 29:ljaf309. doi: 10.1093/bjd/ljaf309. Online ahead of print. PMID 40879371
- [Derived] Chovatiya R, Ribero S, Wollenberg A, Park CO, Silvestre JF, Hong HC, Seneschal J, Saeki H, Thyssen JP, Oland CB, Gjerum L, Maslin D, Blauvelt A. Long-Term Disease Control and Minimal Disease Activity of Head and Neck Atopic Dermatitis in Patients Treated with Tralokinumab up to 4 Years. Am J Clin Dermatol. 2025 Jul;26(4):587-601. doi: 10.1007/s40257-025-00931-1. Epub 2025 Mar 14. PMID 40085349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 309 sites that screened subjects in 11 countries.
Groups:
- Tralokinumab, All Subjects: Week 0: subcutaneous (SC) injection of tralokinumab loading dose.
  From Week 2 up to Week 266*: SC injection of tralokinumab maintenance dose.
  *The length of treatment for each subject will depend on when they enter the trial, and on which parent trial and country they come from.
  Tralokinumab: Human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. Presented as a liquid formulation for subcutaneous injection.
Period: Overall Study
Arm/Group | Tralokinumab, All Subjects
Started | 1672
Completed | 1143
Not Completed | 529
Not completed — Adverse Event | 72
Not completed — Death | 1
Not completed — Lost to Follow-up | 78
Not completed — Withdrawal by Subject | 105
Not completed — Lack of Efficacy | 119
Not completed — Reason unknown | 26
Not completed — COVID_19 pandemic | 4
Not completed — Various reasons | 121
Not completed — Withdrawal by parent/guardian | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tralokinumab, All Subjects
Number analyzed (Participants) | 1672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 103
  Between 18 and 65 years | 1498
  >=65 years | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 709
  Male | 963
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 112
  Not Hispanic or Latino | 1558
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1194
  Black or african american | 120
  Asian | 312
  American indian or alaska native | 2
  Native hawaiian or other pacific islander | 4
  Other | 38
  Missing | 2
Region of Enrollment [Number; unit: participants]
  Canada | 237
  Belgium | 69
  United States | 384
  Czechia | 20
  Japan | 181
  Poland | 228
  Italy | 15
  United Kingdom | 70
  France | 73
  Germany | 268
  Spain | 127
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 77.1 (19.1)
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.3 (10.1)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.52 (6.04)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events From Baseline Through the Last Treatment Visit (up to Week 268)
Time Frame: From Week 0 up to Week 268
Measure: Number; unit: events
Groups:
- Tralokinumab, All Subjects: Week 0: subcutaneous (SC) injection of tralokinumab loading dose.
  From Week 2 up to Week 266: SC injection of tralokinumab maintenance dose.The length of treatment for each subject will depend on when they enter the trial, and on which parent trial and country they come from.
  Tralokinumab: Human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. Presented as a liquid formulation for subcutaneous injection.
Arm/Group | Tralokinumab, All Subjects
Number analyzed (Participants) | 1672
events | 8119

2. Secondary Outcome: Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Weeks 16, 56, 88, 104, 136, 152, 184, 216, and 248
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global atopic dermatitis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: From Week 16 up to Week 248
Population: Modified non-responder analysis with data multiply imputed using a hypothetical strategy. Response is based on observed and multiply imputed data. If a participant permanently discontinued IMP due to lack of efficacy or adverse event before the analyzed visit, they are considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- Tralokinumab, All Subjects: Week 0: subcutaneous (SC) injection of tralokinumab loading dose.
  From Week 2 up to Week 266: SC injection of tralokinumab maintenance dose. The length of treatment for each subject will depend on when they enter the trial, and on which parent trial and country they come from.
  Tralokinumab: Human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. Presented as a liquid formulation for subcutaneous injection.
Arm/Group | Tralokinumab, All Subjects
Number analyzed (Participants) | 1647
percentage of responders
  IGA 0/1 at Week 16 | 47.3 [44.9 to 49.8]
  IGA 0/1 at Week 56 | 48.5 [45.9 to 51.1]
  IGA 0/1 at Week 88 | 48.6 [46.1 to 51.1]
  IGA 0/1 at Week 104 | 47.1 [44.6 to 49.6]
  IGA 0/1 at Week 136 | 48.7 [46.2 to 51.3]
  IGA 0/1 at Week 152 | 46.8 [44.1 to 49.4]
  IGA 0/1 at Week 184 | 46.7 [44.1 to 49.3]
  IGA 0/1 at Week 216 | 47.2 [44.4 to 50.0]
  IGA 0/1 at Week 248 | 46.9 [44.1 to 49.7]

3. Secondary Outcome: At Least 75% Reduction in Eczema Area and Severity Index (EASI75) Relative to Baseline in Parent Trial, at Weeks 16, 56, 88, 104, 136, 152, 184, 216, and 248
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe or more extensive condition.
Time Frame: From Week 16 up to Week 248
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tralokinumab, All Subjects
Number analyzed (Participants) | 1639
percentage of responders
  EASI75 at Week 16 | 77.0 [74.9 to 79.0]
  EASI75 at Week 56 | 75.2 [72.9 to 77.4]
  EASI75 at Week 88 | 75.1 [72.9 to 77.3]
  EASI75 at Week 104 | 74.6 [72.3 to 76.8]
  EASI75 at Week 136 | 74.1 [71.7 to 76.3]
  EASI75 at Week 152 | 73.0 [70.6 to 75.2]
  EASI75 at Week 184 | 72.3 [69.7 to 74.6]
  EASI75 at Week 216 | 72.1 [69.7 to 74.5]
  EASI75 at Week 248 | 71.7 [69.2 to 74.1]

ADVERSE EVENTS:
Time Frame: From baseline up to week 268
Arm/Group | Tralokinumab, All Subjects
All-Cause Mortality (participants affected / at risk) | 1/1672
Serious Adverse Events (participants affected / at risk) | 151/1672
Other Adverse Events (participants affected / at risk) | 924/1672
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab, All Subjects (N=1672)
Angina pectoris (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Atopic cataract (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 3 (3)
Cataract nuclear (Eye disorders) | 1 (1)
Corneal disorder (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2)
Ulcerative keratitis (Eye disorders) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Vogt-Koyanagi-Harada disease (Eye disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Crohn disease (Gastrointestinal disorders) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 4 (4)
Corneal graft rejection (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 5 (5)
Dermatitis infected (Infections and infestations) | 2 (3)
Diverticulitis (Infections and infestations) | 1 (1)
Eczema herpeticum (Infections and infestations) | 3 (3)
Encephalitis herpes (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1)
Herpes zoster pharyngitis (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Medical device site joint infection (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Tonsilitis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Migraine with aura (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (3)
Bladder metaplasia (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 12 (12)
dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1)
Alcohol detoxication (Surgical and medical procedures) | 1 (2)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab, All Subjects (N=1672)
Conjuctivitis (Infections and infestations) | 103 (131)
Covid-19 (Infections and infestations) | 295 (317)
Nasopharyngitis (Infections and infestations) | 372 (599)
Upper respiratory tract infection (Infections and infestations) | 147 (233)
Headache (Nervous system disorders) | 114 (143)
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 351 (620)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03587805/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT03587805/SAP_001.pdf